CLINICAL TRIAL: NCT05849519
Title: Small Sample，Unicentric，Randomized, Controlled Clinical Study of Coenzyme I for Injection in the Treatment of Sudden Sensorineural Hearing Loss
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-KY-004
Record Dates: First submitted 2023-02-16; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-08

CONDITIONS: Sudden Sensorineural Hearing Loss
Keywords: Sudden Sensorineural Hearing Loss; Coenzyme I
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — NAD; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Procedure:Coenzyme I for Injection,5mg，im，qd；Nacl，2ml，im，qd.
  Interventions: Drug: Coenzyme I for Injection + conventional treatment
- Control Group (Other): Procedure: conventional treatment.
  Interventions: Drug: Conventional treatment

INTERVENTIONS:
Drug: Coenzyme I for Injection + conventional treatment — The intervention group used Coenzyme I for injection and conventional treatment for 7 consecutive days
  Arms: Intervention Group
Drug: Conventional treatment — The control group was treated with conventional treatment
  Arms: Control Group

SUMMARY:
Sudden sensorineural hearing loss is one of the most common emergencies in otorhinolaryngology, and its incidence is increasing year by year and tends to be younger. At present, the pathogenesis of sudden deafness is not clear and the individual treatment effects vary significantly. In order to break through this specific treatment bottleneck, this project pioneered the clinical application of the co-regulator nicotinamide adenine dinucleotide (NAD+) in the treatment of sudden deafness. Therefore, this project intends to use pure tone audiometry, speech audiometry, tinnitus disability scale THI, tinnitus subjective visual analog score method VAS, ear fullness subjective visual analog score method VAS for data analysis, and explore the safety of coenzyme I for injection on sudden deafness and efficacy assessment.

DETAILED DESCRIPTION:
The recruited participants were patients with sudden hearing deafness, and the basic demographic data, including name, gender, age, medical history, etc., were collected. According to the inclusion and exclusion criteria, the patients were randomly divided into the experimental group and the control group. The experimental group was given conventional treatment + coenzyme I for injection, and the control group was given conventional treatment for 14 days. Baseline data were collected before treatment, and post-treatment data were collected on 3d, 7d, 14d，1m and 3m of treatment. Baseline data and post-treatment data included pure tone audiometry, speech audiometry, tinnitus THI scale, tinnitus VAS scale, tinnitus Stupid VAS scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18yrs.the 2019 American Sudden Deafness Guidelines are for patients with sudden deafness over 18 years of age;
2. Patients diagnosed with sudden deafness, i.e. unexplained sensorineural hearing loss occurring within 72 hours, with hearing threshold ≥30 in at least 3 consecutive frequencies, refer to the 2019 American Sudden Deafness Guidelines;
3. Unilateral sudden deafness;
4. Within 1 week of the onset of sudden deafness, no treatment in another hospital/our hospital;
5. No major neurological disease, serious systemic disease, family genetic history, major mental illness;
6. Informed and agreed to join the experiment, no plan to move out or go out within 1 month.

Exclusion Criteria:

1. Other diseases such as acoustic neuroma diagnosed by imaging;
2. Those who cannot tolerate NAD+;
3. pregnant；
4. Any other circumstances that the investigator believes should be excluded from this study；
5. Do not agree to join the experiment, plan to move out or go out within 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-02-16 (Estimated); Study Completion 2024-02-16 (Estimated)

PRIMARY OUTCOMES:
Pure Tone Average(PTA) | Baseline, before treatment
  Pure tone audiometry is the most basic and preferred hearing test method, which can qualitatively and quantitatively diagnose hearing loss, can reflect the entire auditory conduction pathway from the external ear to the auditory center, and is currently one of the subjective behavioral hearing tests that can accurately reflect hearing acuity. Includes pure tone air conduction hearing threshold test and pure tone bone hearing threshold test.
Pure Tone Average(PTA) | Treatment day 3
  Pure tone audiometry is the most basic and preferred hearing test method, which can qualitatively and quantitatively diagnose hearing loss, can reflect the entire auditory conduction pathway from the external ear to the auditory center, and is currently one of the subjective behavioral hearing tests that can accurately reflect hearing acuity. Includes pure tone air conduction hearing threshold test and pure tone bone hearing threshold test.
Pure Tone Average(PTA) | Treatment day 7
  Pure tone audiometry is the most basic and preferred hearing test method, which can qualitatively and quantitatively diagnose hearing loss, can reflect the entire auditory conduction pathway from the external ear to the auditory center, and is currently one of the subjective behavioral hearing tests that can accurately reflect hearing acuity. Includes pure tone air conduction hearing threshold test and pure tone bone hearing threshold test.
Pure Tone Average(PTA) | Treatment day 14
  Pure tone audiometry is the most basic and preferred hearing test method, which can qualitatively and quantitatively diagnose hearing loss, can reflect the entire auditory conduction pathway from the external ear to the auditory center, and is currently one of the subjective behavioral hearing tests that can accurately reflect hearing acuity. Includes pure tone air conduction hearing threshold test and pure tone bone hearing threshold test.
Pure Tone Average(PTA) | Treatment day 30
  Pure tone audiometry is the most basic and preferred hearing test method, which can qualitatively and quantitatively diagnose hearing loss, can reflect the entire auditory conduction pathway from the external ear to the auditory center, and is currently one of the subjective behavioral hearing tests that can accurately reflect hearing acuity. Includes pure tone air conduction hearing threshold test and pure tone bone hearing threshold test.
Pure Tone Average(PTA) | Treatment day 90
  Pure tone audiometry is the most basic and preferred hearing test method, which can qualitatively and quantitatively diagnose hearing loss, can reflect the entire auditory conduction pathway from the external ear to the auditory center, and is currently one of the subjective behavioral hearing tests that can accurately reflect hearing acuity. Includes pure tone air conduction hearing threshold test and pure tone bone hearing threshold test.

SECONDARY OUTCOMES:
Speech Recognition Rate | Baseline, before treatment
  The speech recognition rate is the percentage (%) of speech which can be heard correctly in the audiometric vocabulary list, and the curve is drawn according to the (%) understood by different sound intensity levels, that is, the speech audiogram.
Speech Recognition Rate | Treatment day 3
  The speech recognition rate is the percentage (%) of speech which can be heard correctly in the audiometric vocabulary list, and the curve is drawn according to the (%) understood by different sound intensity levels, that is, the speech audiogram.
Speech Recognition Rate | Treatment day 7
  The speech recognition rate is the percentage (%) of speech which can be heard correctly in the audiometric vocabulary list, and the curve is drawn according to the (%) understood by different sound intensity levels, that is, the speech audiogram.
Speech Recognition Rate | Treatment day 14
  The speech recognition rate is the percentage (%) of speech which can be heard correctly in the audiometric vocabulary list, and the curve is drawn according to the (%) understood by different sound intensity levels, that is, the speech audiogram.
Speech Recognition Rate | Treatment day 30
  The speech recognition rate is the percentage (%) of speech which can be heard correctly in the audiometric vocabulary list, and the curve is drawn according to the (%) understood by different sound intensity levels, that is, the speech audiogram.
Speech Recognition Rate | Treatment day 90
  The speech recognition rate is the percentage (%) of speech which can be heard correctly in the audiometric vocabulary list, and the curve is drawn according to the (%) understood by different sound intensity levels, that is, the speech audiogram.
Tinnitus Handicap Inventory | Baseline, before treatment
  The Tinnitus Handicap Inventory (THI) is a tool to measure the impact of tinnitus on daily life.
  Yes (always has): 4 points; Sometimes (intermittent presence): 2 points.None: 0 points; None:0 points. Divide tinnitus into grade 5 I (mild), THI score 1~16 divide; Grade 2 (mild), THI score 18~36 points; Level 3 (moderate), THI score 38~56 points; Level 4 (severe), THI score 58~76 points; Level 5 (catastrophic), THI score 78~100 points.
Tinnitus Handicap Inventory | Treatment day 3
  The Tinnitus Handicap Inventory (THI) is a tool to measure the impact of tinnitus on daily life.
  Yes (always has): 4 points; Sometimes (intermittent presence): 2 points.None: 0 points; None:0 points. Divide tinnitus into grade 5 I (mild), THI score 1~16 divide; Grade 2 (mild), THI score 18~36 points; Level 3 (moderate), THI score 38~56 points; Level 4 (severe), THI score 58~76 points; Level 5 (catastrophic), THI score 78~100 points.
Tinnitus Handicap Inventory | Treatment day 7
  The Tinnitus Handicap Inventory (THI) is a tool to measure the impact of tinnitus on daily life.
  Yes (always has): 4 points; Sometimes (intermittent presence): 2 points.None: 0 points; None:0 points. Divide tinnitus into grade 5 I (mild), THI score 1~16 divide; Grade 2 (mild), THI score 18~36 points; Level 3 (moderate), THI score 38~56 points; Level 4 (severe), THI score 58~76 points; Level 5 (catastrophic), THI score 78~100 points.
Tinnitus Handicap Inventory | Treatment day 14
  The Tinnitus Handicap Inventory (THI) is a tool to measure the impact of tinnitus on daily life.
  Yes (always has): 4 points; Sometimes (intermittent presence): 2 points.None: 0 points; None:0 points. Divide tinnitus into grade 5 I (mild), THI score 1~16 divide; Grade 2 (mild), THI score 18~36 points; Level 3 (moderate), THI score 38~56 points; Level 4 (severe), THI score 58~76 points; Level 5 (catastrophic), THI score 78~100 points.
Tinnitus Handicap Inventory | Treatment day 30
  The Tinnitus Handicap Inventory (THI) is a tool to measure the impact of tinnitus on daily life.
  Yes (always has): 4 points; Sometimes (intermittent presence): 2 points.None: 0 points; None:0 points. Divide tinnitus into grade 5 I (mild), THI score 1~16 divide; Grade 2 (mild), THI score 18~36 points; Level 3 (moderate), THI score 38~56 points; Level 4 (severe), THI score 58~76 points; Level 5 (catastrophic), THI score 78~100 points.
Tinnitus Handicap Inventory | Treatment day 90
  The Tinnitus Handicap Inventory (THI) is a tool to measure the impact of tinnitus on daily life.
  Yes (always has): 4 points; Sometimes (intermittent presence): 2 points.None: 0 points; None:0 points. Divide tinnitus into grade 5 I (mild), THI score 1~16 divide; Grade 2 (mild), THI score 18~36 points; Level 3 (moderate), THI score 38~56 points; Level 4 (severe), THI score 58~76 points; Level 5 (catastrophic), THI score 78~100 points.
Visual Analogue Scale of Tinnitus | Baseline, before treatment
  VAS (Visual Analogue Scale) is a tool to detect changes in the subjective loudness of tinnitus. 0 represents no tinnitus loudness at all, 10 represents the presence of extremely severe loudness, and the middle represents different degrees of tinnitus loudness.
Visual Analogue Scale of Tinnitus | Treatment day 3
  VAS (Visual Analogue Scale) is a tool to detect changes in the subjective loudness of tinnitus. 0 represents no tinnitus loudness at all, 10 represents the presence of extremely severe loudness, and the middle represents different degrees of tinnitus loudness.
Visual Analogue Scale of Tinnitus | Treatment day 7
  VAS (Visual Analogue Scale) is a tool to detect changes in the subjective loudness of tinnitus. 0 represents no tinnitus loudness at all, 10 represents the presence of extremely severe loudness, and the middle represents different degrees of tinnitus loudness.
Visual Analogue Scale of Tinnitus | Treatment day 14
  VAS (Visual Analogue Scale) is a tool to detect changes in the subjective loudness of tinnitus. 0 represents no tinnitus loudness at all, 10 represents the presence of extremely severe loudness, and the middle represents different degrees of tinnitus loudness.
Visual Analogue Scale of Tinnitus | Treatment day 30
  VAS (Visual Analogue Scale) is a tool to detect changes in the subjective loudness of tinnitus. 0 represents no tinnitus loudness at all, 10 represents the presence of extremely severe loudness, and the middle represents different degrees of tinnitus loudness.
Visual Analogue Scale of Tinnitus | Treatment day 90
  VAS (Visual Analogue Scale) is a tool to detect changes in the subjective loudness of tinnitus. 0 represents no tinnitus loudness at all, 10 represents the presence of extremely severe loudness, and the middle represents different degrees of tinnitus loudness.
Severity of ear fullness | Baseline, before treatment
  Visual Analogue Scale(VAS).0 represents no ear stuffiness at all, 10 represents the presence of extremely severe ear stuffiness, and the middle represents different degrees of ear stuffiness.
Severity of ear fullness | Treatment day 3
  Visual Analogue Scale(VAS).0 represents no ear stuffiness at all, 10 represents the presence of extremely severe ear stuffiness, and the middle represents different degrees of ear stuffiness.
Severity of ear fullness | Treatment day 7
  Visual Analogue Scale(VAS).0 represents no ear stuffiness at all, 10 represents the presence of extremely severe ear stuffiness, and the middle represents different degrees of ear stuffiness.
Severity of ear fullness | Treatment day 14
  Visual Analogue Scale(VAS).0 represents no ear stuffiness at all, 10 represents the presence of extremely severe ear stuffiness, and the middle represents different degrees of ear stuffiness.
Severity of ear fullness | Treatment day 30
  Visual Analogue Scale(VAS).0 represents no ear stuffiness at all, 10 represents the presence of extremely severe ear stuffiness, and the middle represents different degrees of ear stuffiness.
Severity of ear fullness | Treatment day 90
  Visual Analogue Scale(VAS).0 represents no ear stuffiness at all, 10 represents the presence of extremely severe ear stuffiness, and the middle represents different degrees of ear stuffiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China